CLINICAL TRIAL: NCT07127705
Title: Rapid Response of Stem Cells and Immune Cells for Efficacy: An Acute Randomized Double-blind Placebo-controlled Cross-over Trial
Brief Title: Rapid Response of Stem Cells and Immune Cells for Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Collaborators: Applied Food Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 186-006
Record Dates: First submitted 2025-05-19; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Stem Cell Surveillance
MeSH Terms: interventions — Asian ginseng; olive extract; potassium hydrogen glucarate

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, double-blinded, cross-over study design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crossover group 1, randomized (Experimental): Crossover study: Participants consume a test product on each of the five clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 4 active test products versus placebo over 5 weeks. The order of interventions for this group is A, C, B, D, E.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Chaga Mushroom; Dietary Supplement: Ginseng extract; Dietary Supplement: Olive extract; Dietary Supplement: Potassium Hydrogen Glucarate
- Crossover group 2, randomized (Experimental): Crossover study: Participants consume a test product on each of the five clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 4 active test products versus placebo over 5 weeks. The order of interventions for this group is E, A, C, B, D.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Chaga Mushroom; Dietary Supplement: Ginseng extract; Dietary Supplement: Olive extract; Dietary Supplement: Potassium Hydrogen Glucarate
- Crossover group 3, randomized (Experimental): Crossover study: Participants consume a test product on each of the five clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 4 active test products versus placebo over 5 weeks. The order of interventions for this group is D, E, A, C, B.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Chaga Mushroom; Dietary Supplement: Ginseng extract; Dietary Supplement: Olive extract; Dietary Supplement: Potassium Hydrogen Glucarate
- Crossover group 4, randomized (Experimental): Crossover study: Participants consume a test product on each of the five clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 4 active test products versus placebo over 5 weeks. The order of interventions for this group is B, C, D, A, E.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Chaga Mushroom; Dietary Supplement: Ginseng extract; Dietary Supplement: Olive extract; Dietary Supplement: Potassium Hydrogen Glucarate

INTERVENTIONS:
Dietary Supplement: Placebo — 2 capsules
Dietary Supplement: Chaga Mushroom — 2 capsules
Dietary Supplement: Ginseng extract — 2 capsules
Dietary Supplement: Olive extract — 2 capsules
Dietary Supplement: Potassium Hydrogen Glucarate — 2 capsules

SUMMARY:
The goal for this clinical trial is to compare rapid effects of four products on stem cells, immune activation, and mitochondrial function. A double-blind, placebo-controlled, cross-over study design will be used.

DETAILED DESCRIPTION:
This clinical trial aims at documenting acute effects of consuming four products through evaluation of stem cell surveillance and mitochondrial resilience.

Data on stem cell trafficking will be collected. The testing will show whether consuming the products leads to a rapid change in stem cell surveillance. Data on cellular energy production and mitochondrial resilience in white blood cells under oxidative and inflammatory stress ex vivo will be collected. This testing will show whether consuming the test products leads to support of energy production within mitochondria, under normal and stressed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18 - 75 years (inclusive);
* BMI between 18.0 and 34.9 (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:

  * Maintaining a consistent diet and lifestyle routine throughout the study,
  * Consistent habit of bland breakfasts on days of clinic visits,
  * Abstaining from exercising and nutritional supplements on the morning of a study visit,
  * Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
  * Abstaining from music, candy, gum, computer/cell phone use (airplane mode is allowed), during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-08-27 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Stem cell trafficking | Baseline. 1 hour, 2 hours, and 3 hours after ingestion of study drug
  Changes to the number of stem cells in the blood circulation (number of cells per mL blood).
  Data is collected on the following types of stem cells: CD45dimCD34+CD309+, CD45dimCD34+CD309-, CD31++CD34-, CD45-CD90+.

SECONDARY OUTCOMES:
Mitochondrial volume per cell | Baseline. 1 hour, 2 hours, 3 and hours after ingestion of study drug
  Mitochondrial volume per cell under unstressed, oxidative stress, and inflammatory stress ex vivo. White blood cells are purified and cultured ex vivo in unstressed versus inflamed culture conditions. The mitochondrial reporter dye MitoTracker is used to obtain relative measures of mitochondrial volume per cell using flow cytometry, where the mean fluorescence intensity (MFI) is quantified on lymphocytes, monocytes, and PMN cells.
Mitochondrial membrane potential per cell | Baseline. 1 hour, 2 hours, and 3 hours after ingestion of study drug
  Cellular energy production under unstressed, oxidative stress, and inflammatory stress ex vivo. White blood cells are purified and cultured ex vivo in unstressed versus inflamed culture conditions. The mitochondrial reporter dye JC-1 is a fluorescent cationic dye used to obtain relative measures of mitochondrial membrane potential per cells, using flow cytometry, where the mean fluorescence intensity (MFI) is quantified on lymphocytes, monocytes, and PMN cells.

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No